CLINICAL TRIAL: NCT05245071
Title: Open-label, Phase 2 Study, Evaluating the Efficacy and Safety of Tusamitamab Ravtansine in Non-squamous Non-small-cell Lung Cancer (NSQ NSCLC) Participants With Negative or Moderate CEACAM5 Expression Tumors and High Circulating CEA
Brief Title: Tusamitamab Ravtansine in NSQ NSCLC Participants With Negative or Moderate CEACAM5 Expression Tumors and High Circulating CEA
Acronym: CARMEN-LC06
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision, the decision is not related to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT17241; U1111-1264-2828 (Registry Identifier: ICTRP); 2021-004423-32 (EudraCT Number)
Record Dates: First submitted 2022-02-09; First posted 2022-02-17 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — tusamitamab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tusamitamab ravtansine (Experimental): Tusamitamab ravtansine dose will be administered on Day 1 via IV infusion and repeated once every 2 weeks. The duration of 1 cycle will be 14 days (1 administration of tusamitamab ravtansine per cycle).
  Interventions: Drug: Tusamitamab ravtansine

INTERVENTIONS:
Drug: Tusamitamab ravtansine — Pharmaceutical Form: Concentrate for solution Route of Administration: Intravenous infusion
  Other Names: SAR408701

SUMMARY:
This is an open label single group, Phase 2, 1-arm study for treatment to evaluate efficacy, safety, and Pharmacokinetic (PK) of tusamitamab ravtansine in nonsquamous non-small-cell-lung-cancer (NSQ NSCLC) participants with negative or moderate CEACAM5 expression tumors and high circulating carcinoembryonic antigen (CEA).

Participants who will be enrolled, will receive tusamitamab ravtansine as monotherapy every two weeks (Q2W) until disease progression, unacceptable adverse event (AE), initiation of a new anticancer therapy, or the participant's or investigator's decision to stop the treatment, whichever comes first. A total of approximately 38 participants are planned to be treated.

DETAILED DESCRIPTION:
40 weeks (up to 4 weeks for screening, a median of 24 weeks for treatment, and a median of 12 weeks for end of treatment assessments and the safety follow-up visit).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of NSQ NSCLC metastatic disease at study entry; progression after platinum-based chemotherapy and immune checkpoint inhibitor.
* Participants with moderate or negative CEACAM5 expression as demonstrated prospectively by central laboratory via immune histochemistry (ICH) and high circulating CEA levels (≥100 ng/mL). Moderate CEACAM5 expression is defined as intensity ≥ 2 + in ≥ 1% and <50 % of tumor cells. Negative CEACAM5 expression is defined as intensity of 1 + whatever the percentage of stained tumor cells or <1% of tumor cells.
* At least one measurable lesion by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Women of childbearing potential or male patient with women of childbearing potential who agree to use highly effective method of birth control.

Exclusion Criteria:

* Patients with untreated brain metastases or history of leptomeningeal disease.
* History within the last 3 years of an invasive malignancy other than the one treated in this study, with the exception of resected/ablated basal or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix, or other local tumors considered cured by local treatment.
* History of known uncontrolled infection with human immunodeficiency virus (HIV), or unresolved viral hepatitis
* Significant concomitant illness that could impair the participation in the study or interpretation of the results or any major surgery with 3 weeks prior treatment administration
* Nonresolution of any prior treatment-related toxicity to <Grade 2 according to NCI CTCAE v5.0, with the exception of alopecia, vitiligo, or active thyroiditis controlled with hormone replacement therapy.
* Previous history of and/or unresolved corneal disorders. The use of contact lenses is not permitted.
* Prior treatment with maytansinoid derivatives (DM1 or DM4 antibody drug conjugate) or any drug targeting CEACAM5.
* Concurrent treatment with any other anticancer therapy
* Poor bone marrow, liver or kidney functions.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (35):
- United States (2):
  - Roswell Park Cancer Institute Site Number : 8400004, Buffalo, New York
  - Renovatio Clinical Site Number : 8400003, El Paso, Texas
- Belgium (3):
  - Investigational Site Number : 0560003, Edegem
  - Investigational Site Number : 0560001, Leuven
  - Investigational Site Number : 0560002, Liège
- France (8):
  - Investigational Site Number : 2500003, Bordeaux
  - Investigational Site Number : 2500001, Créteil
  - Investigational Site Number : 2500007, Marseille
  - Investigational Site Number : 2500005, Montpellier
  - Investigational Site Number : 2500002, Rennes
  - Investigational Site Number : 2500006, Saint-Herblain
  - Investigational Site Number : 2500008, Saint-Mandé
  - Investigational Site Number : 2500009, Villejuif
- Italy (4):
  - Investigational Site Number : 3800003, Ravenna, Emilia-Romagna
  - Investigational Site Number : 3800004, Aviano (PN), Friuli Venezia Giulia
  - Investigational Site Number : 3800001, Rozzano, Lombardy
  - Investigational Site Number : 3800002, Milan
- Japan (4):
  - Investigational Site Number : 3920002, Nagoya, Aichi-ken
  - Investigational Site Number : 3920001, Sapporo, Hokkaido
  - Investigational Site Number : 3920005, Hirakata-shi, Osaka
  - Investigational Site Number : 3920003, Sunto Gun, Shizuoka
- Spain (9):
  - Investigational Site Number : 7240004, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240006, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240008, Majadahonda, Madrid
  - Investigational Site Number : 7240002, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240009, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240003, Málaga
  - Investigational Site Number : 7240005, Seville
  - Investigational Site Number : 7240007, Valencia
- Turkey (Türkiye) (5):
  - Investigational Site Number : 7920002, Adana
  - Investigational Site Number : 7920005, Ankara
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920004, Istanbul
  - Investigational Site Number : 7920001, Malatya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 35 investigational sites in 7 countries. A total of 30 participants were screened from 01-Jun-2022 to 01-Dec-2023 of which 8 were screen failures due to not meeting eligibility criteria. The study was terminated as per Sponsor decision and not related to any safety concern.
Pre-assignment Details: A total of 22 participants were enrolled in the study. Note: Reason for not completed = Reason for permanent full study intervention discontinuation.
Groups:
- Tusamitamab Ravtansine 100 Milligrams Per Meter Square (mg/m^2): Participants received tusamitamab ravtansine 100 mg/m^2 via intravenous (IV) infusion every 2 weeks (Q2W) until disease progression, unacceptable adverse event (AE), death, initiation of a new anticancer therapy, or the participant's or investigator's decision to stop the treatment.
Period: Overall Study
Arm/Group | Tusamitamab Ravtansine 100 Milligrams Per Meter Square (mg/m^2)
Started | 22
Completed | 0
Not Completed | 22
Not completed — Progressive disease | 18
Not completed — Adverse event not related to Coronavirus Disease 2019 | 2
Not completed — Not related to Coronavirus Disease 2019 | 2

BASELINE CHARACTERISTICS:
Population: All-treated population included all enrolled participants exposed to the study treatment, regardless of the amount of treatment administered.
Groups:
- Tusamitamab Ravtansine 100 mg/m^2: Participants received tusamitamab ravtansine 100 mg/m^2 via IV infusion Q2W until disease progression, unacceptable AE, death, initiation of a new anticancer therapy, or the participant's or investigator's decision to stop the treatment.
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as percentage of participants with confirmed complete response (CR) or partial response (PR) as best overall response (BOR) determined per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. The CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm). The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Tumor assessments performed at baseline, and every 8 weeks +/-7 days thereafter, approximately 46 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2
Number analyzed (Participants) | 22
percentage of participants | 9.1 [1.12 to 29.16]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death or was life-threatening or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent disability/incapacity or congenital anomaly/birth defect or was a suspected transmission of any infectious agent via an authorized medicinal product. TEAE was defined as AEs that developed, worsened, or became serious during the treatment-emergent period.
Time Frame: From the first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment, approximately 84 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2
Number analyzed (Participants) | 22
Participants
  Any TEAEs | 21
  Any TESAEs | 7

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: The PFS was defined as the time from the first study treatment administration to the date of the first documented progressive disease (PD) or death due to any cause, whichever came first as per RECIST v1.1. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions was also considered progression.
Time Frame: Tumor assessments performed at baseline, and every 8 weeks +/-7 days thereafter, approximately 46 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2
Number analyzed (Participants) | 22
months | 1.87 [1.676 to 3.614]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR was defined as the percentage of participants who achieved confirmed CR, PR or stable disease (SD) as BOR as per RECIST v1.1. The CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. The PR was defined as at least a 30%decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD was defined as neither sufficient shrinkage from the baseline study to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on the study.
Time Frame: Tumor assessments performed at baseline, and every 8 weeks +/-7 days thereafter, approximately 46 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2
Number analyzed (Participants) | 22
percentage of participants | 36.4 [17.20 to 59.34]

5. Secondary Outcome: Duration of Response (DOR)
Description: The DOR was defined as the time from first documented evidence of CR or PR until PD determined per RECIST v1.1 or death from any cause, whichever occurred first. The CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Tumor assessments performed at baseline, and every 8 weeks +/-7 days thereafter, approximately 46 weeks
Population: All-treated population included all enrolled participants exposed to the study treatment, regardless of the amount of treatment administered. Only responders (those participants with confirmed CR or PR) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2
Number analyzed (Participants) | 2
months | NA [NA to NA] — NA indicates that data was not estimable due to insufficient number of participants with events until primary completion date of 06-Mar-2024.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment, approximately 84 weeks. All-cause mortality (death) was assessed from signing of the informed consent form (Day -28) to study termination, up to 129 weeks.
Description: Analysis was performed on all-treated population.
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2
All-Cause Mortality (participants affected / at risk) | 13/22
Serious Adverse Events (participants affected / at risk) | 7/22
Other Adverse Events (participants affected / at risk) | 18/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tusamitamab Ravtansine 100 mg/m^2 (N=22)
Pneumonia (Infections and infestations) | 2 (3)
Epilepsy (Nervous system disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Right Ventricular Failure (Cardiac disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tusamitamab Ravtansine 100 mg/m^2 (N=22)
Decreased Appetite (Metabolism and nutrition disorders) | 9 (10)
Keratitis (Eye disorders) | 3 (6)
Keratopathy (Eye disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (7)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Renal Failure (Renal and urinary disorders) | 2 (2)
Asthenia (General disorders) | 6 (7)
Fatigue (General disorders) | 3 (3)
Non-Cardiac Chest Pain (General disorders) | 3 (3)
Oedema Peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Weight Decreased (Investigations) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was terminated as per Sponsor decision and not related to any safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT05245071/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT05245071/SAP_001.pdf